CLINICAL TRIAL: NCT00672477
Title: A Randomized, Double-Blind, Placebo-Controlled Study Of A Fixed Dose Of Subcutaneous Methylnaltrexone In Adults With Advanced Illness And Opioid-Induced Constipation: Efficacy, Safety, And Additional Health Outcomes
Brief Title: Study Evaluating Subcutaneous Methylnaltrexone For Treatment Of Opioid-Induced Constipation In Patients With Advanced Illness
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Collaborators: Progenics Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3200K1-4000; B2541005
Record Dates: First submitted 2008-05-02; First posted 2008-05-06 (Estimated); Results first posted 2018-03-08 (Actual); Last update posted 2018-03-08 (Actual); Status verified 2018-02

CONDITIONS: Opioid-Induced Constipation
Keywords: opioid-induced constipation
MeSH Terms: conditions — Opioid-Induced Constipation | interventions — methylnaltrexone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Methylnaltrexone (Experimental): Methylnaltrexone subcutaneously every other day for 14 days (ie, 7 doses). Subjects received 0.6 mL (12 mg) every other day if weight ≥ 62kg; or 0.4 mL (8 mg) every other day if weight between 38 and <62 kg. Subjects with impaired kidney function received reduced doses according to instructions in the Relistor prescribing information.
  Interventions: Drug: Methylnaltrexone
- Placebo (Placebo Comparator): Placebo subcutaneously every other day for 14 days (ie, 7 doses). Subjects received 0.6 mL every other day if weight ≥ 62kg; or 0.4 mL every other day if weight between 38 and < 62 kg. Subjects with impaired kidney function received reduced volumes of placebo solution to match the volumes used in the experimental group.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methylnaltrexone
  Other Names: MOA-728; Relistor
  Arms: Methylnaltrexone
Drug: Placebo
  Other Names: Control
  Arms: Placebo

SUMMARY:
This study will evaluate the safety and efficacy of methylnaltrexone administered as subcutaneous injections in subjects who have opioid-induced constipation and an advanced illness. The hypothesis is that methylnaltrexone will be safe and effective in relieving opioid-induced constipation in these subjects.

ELIGIBILITY:
Inclusion Criteria:

* Is an adult 18 years of age or older
* Has a diagnosis of advanced illness (ie, a terminal illness such as incurable cancer or other end-stage disease)
* Has a life expectancy of at least 1 month.
* Is receiving opioids on a regular schedule (not just as-needed or rescue doses) for the control of pain or discomfort for at least 2 weeks before the first dose of study drug.
* Has constipation that is caused by opioid medications.

Exclusion Criteria:

* Has a known or suspected allergy to methylnaltrexone or other similar compounds (e.g. naltrexone or naloxone).
* Has a known or suspected mechanical gastrointestinal obstruction.
* Has any potential nonopioid cause of bowel dysfunction that might be a major contributor to the constipation.
* Has any other clinically important abnormalities as determined by the investigator that may interfere with his or her participation in or compliance with the study.
* Receiving opioid antagonist or partial antagonist products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2008-06; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Enoch Bortey, Study Director — Bausch Health Americas, Inc.
Locations (54):
- United States (26):
  - Salix Investigational Site, Mobile, Alabama
  - Salix Investigational Site, Laguna Hills, California
  - Salix Investigational Site, Lancaster, California
  - Salix Investigational Site, Aurora, Colorado
  - Salix Investigational Site, Auburndale, Florida
  - Salix Investigational Site, Hudson, Florida
  - Salix Investigational Site, Lakeland, Florida
  - Salix Investigational Site, Miami Springs, Florida
  - Salix Investigational Site, Ruskin, Florida
  - Salix Investigational Site, Sebring, Florida
  - Salix Investigational Site, Tampa, Florida
  - Salix Investigational Site, Temple Terrace, Florida
  - Salix Investigational Site, West Palm Beach, Florida
  - Salix Investigational Site, Orange, New Jersey
  - Salix Investigational Site, Albuquerque, New Mexico
  - Salix Investigational Site, Flat Rock, North Carolina
  - Salix Investigational Site, Winston-Salem, North Carolina
  - Salix Investigational Site, Cleveland, Ohio
  - Salix Investigational Site, Philadelphia, Pennsylvania
  - Salix Investigational Site, Austin, Texas
  - Salix Investigational Site, Houston, Texas
  - Salix Investigational Site, American Fork, Utah
  - Salix Investigational Site, Orem, Utah
  - Salix Investigational Site, Provo, Utah
  - Salix Investigational Site, Salt Lake City, Utah
  - Salix Investigational Site, Madison, Wisconsin
- Australia (3):
  - Salix Investigational Site, Darlinghurst, New South Wales
  - Salix Investigational Site, Coburg, Victoria
  - Salix Investigational Site, East Melbourne, Victoria
- Salix Investigational Site, Leuven, Belgium
- Brazil (2):
  - Salix Investigational Site, Liberdade, São Paulo
  - Salix Investigational Site, São Paulo, São Paulo
- Canada (5):
  - Salix Investigational Site, Edmonton, Alberta
  - Salix Investigational Site, Winnipeg, Manitoba
  - Salix Investigational Site, Hamilton, Ontario
  - Salix Investigational Site, Montreal, Quebec
  - Salix Investigational Site, Québec, Quebec
- France (5):
  - Salix Investigational Site, Besançon
  - Salix Investigational Site, Bordeaux
  - Salix Investigational Site, Grenoble
  - Salix Investigational Site, Montpellier
  - Salix Investigational Site, Villejuif
- Germany (3):
  - Salix Investigational Site, Aachen
  - Salix Investigational Site, Berlin
  - Salix Investigational Site, München
- Italy (2):
  - Salix Investigational Site, L’Aquila
  - Salix Investigational Site, Milan
- Pfizer Investigational Site, Mexico City DF, Mexico
- Spain (3):
  - Salix Investigational Site, Barcelona
  - Salix Investigational Site, L'Hospitalet de Llobregat
  - Salix Investigational Site, Seville
- Sweden (2):
  - Salix Investigational Site, Kungsbacka
  - Salix Investigational Site, Norrköping
- Salix Investigational Site, Cheltenham, Gloucestershire, United Kingdom

REFERENCES:
- [Derived] Liao SS, Slatkin NE, Stambler N. The Influence of Age on Central Effects of Methylnaltrexone in Patients with Opioid-Induced Constipation. Drugs Aging. 2021 Jun;38(6):503-511. doi: 10.1007/s40266-021-00850-w. Epub 2021 Mar 31. PMID 33788162
- [Derived] Janku F, Johnson LK, Karp DD, Atkins JT, Singleton PA, Moss J. Treatment with methylnaltrexone is associated with increased survival in patients with advanced cancer. Ann Oncol. 2016 Nov;27(11):2032-2038. doi: 10.1093/annonc/mdw317. Epub 2016 Aug 29. PMID 27573565

RESULTS

PARTICIPANT FLOW:
Groups:
- Methylnaltrexone Bromide: Methylnaltrexone bromide: Methylnaltrexone subcutaneously every other day for 14 days (ie, 7 doses).
- Placebo: Placebo: Placebo subcutaneously every other day for 14 days (ie, 7 doses).
Period: Overall Study
Arm/Group | Methylnaltrexone Bromide | Placebo
Started | 116 (120 subjects were randomized to this group, but only 116 subjects received study drug.) | 114 (117 subjects were randomized to this group, but only 114 subjects received study drug.)
Completed | 89 (One subject had missing data as reason for study termination - not counted as early termination.) | 88
Not Completed | 27 | 26
Not completed — Adverse Event | 10 | 7
Not completed — Death | 7 | 11
Not completed — Physician Decision | 2 | 0
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Lack of Efficacy | 1 | 1
Not completed — no study drug for low GFR, health cond. | 1 | 3

BASELINE CHARACTERISTICS:
Population: The analysis population included subjects who received ≥ 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Methylnaltrexone Bromide | Placebo | Total
Number analyzed (Participants) | 116 | 114 | 230
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 60 | 57 | 117
  >=65 years | 56 | 57 | 113
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.31 (12.92) | 65.67 (12.97) | 65.49 (12.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 58 | 114
  Male | 60 | 56 | 116
Underlying Advanced Illness [Number; unit: participants]
  Cancer | 79 | 73 | 152
  Pulmonary disease (other than malignancy) | 14 | 13 | 27
  Cardiovascular disease | 13 | 11 | 24
  Neurologic disease | 4 | 3 | 7
  Other | 6 | 14 | 20
Weight [Number; unit: participants]
  < 62 kg | 45 | 41 | 86
  ≥ 62 kg | 71 | 73 | 144
Glomerular filtration rate [Number; unit: participants]
  < 30 mL/min/1.73 m^2 | 3 | 3 | 6
  ≥ 30 mL/min/1.73 m^2 | 110 | 108 | 218
  Missing | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Subjects Who Have a Rescue-free Laxation Response Within 4 Hours After at Least 2 of the First 4 Doses
Description: This outcome measures the proportion of subjects who had a rescue-free laxation (ie, bowel movement) within 4 hours after at least 2 of the first 4 doses of study drug. A "rescue free" laxation was defined as a laxation without use of any rescue medication or rescue procedures within 4 hours prior to the laxation.
Time Frame: 7 days
Population: The analysis population included subjects who received ≥ 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Methylnaltrexone Bromide | Placebo
Number analyzed (Participants) | 116 | 114
percentage of participants | 62.9 [53.5 to 71.7] | 9.6 [4.9 to 16.6]
Statistical Analysis 1: Comparison: Methylnaltrexone Bromide vs Placebo; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel

2. Secondary Outcome: Time to First Rescue-free Laxation (Following the First Dose of Study Drug).
Description: This outcome measures the time from first dose of study drug to the first rescue-free laxation (ie, bowel movement). A "rescue free" laxation was defined as a laxation without use of any rescue medication or rescue procedures within 4 hours prior to the laxation.
Time Frame: 14 days
Population: The analysis population included subjects who received ≥ 1 dose of study drug.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Methylnaltrexone Bromide | Placebo
Number analyzed (Participants) | 116 | 114
hours | 0.79 [0.38 to 6.17] | 23.58 [6.75 to 47.00]
Statistical Analysis 1: Comparison: Methylnaltrexone Bromide vs Placebo; Test type: Superiority or Other; p < 0.0001, Log Rank

ADVERSE EVENTS:
Time Frame: 14 days
Description: Adverse events were collected by non-systematic (patient reports) and systematic methods (investigator examinations and lab tests). For both adverse events tables, a subject reporting more than one adverse event for a particular MedDRA preferred term or system organ class was counted only once for that MedDRA preferred term or system organ class.
Arm/Group | Methylnaltrexone Bromide | Placebo
Serious Adverse Events (participants affected / at risk) | 14/116 | 24/114
Other Adverse Events (participants affected / at risk) | 66/116 | 52/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Methylnaltrexone Bromide (N=116) | Placebo (N=114)
Anemia (Blood and lymphatic system disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Disease progression (General disorders) | 9 | 14
Fall (Injury, poisoning and procedural complications) | 0 | 2
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Spinal cord compression (Nervous system disorders) | 0 | 2
Delirium (Psychiatric disorders) | 0 | 1
Disorientation (Psychiatric disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Gastric ulcer perforation (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Methylnaltrexone Bromide (N=116) | Placebo (N=114)
Abdominal pain (Gastrointestinal disorders) | 39 | 19
Diarrhea (Gastrointestinal disorders) | 9 | 15
Flatulence (Gastrointestinal disorders) | 8 | 5
Nausea (Gastrointestinal disorders) | 13 | 17
Vomiting (Gastrointestinal disorders) | 5 | 10
Edema peripheral (General disorders) | 7 | 4
Fall (Injury, poisoning and procedural complications) | 9 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 3
Confusional state (Psychiatric disorders) | 7 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less